CLINICAL TRIAL: NCT06210048
Title: Investigation of Sacroiliac Joint Dysfunction and Spinal Mobility in Women With Primary Dysmenorrhoea
Brief Title: Sacroiliac Joint Dysfunction and Spinal Mobility in Women With Primary Dysmenorrhoea
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ömer Osman Pala, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-OOP-2
Record Dates: First submitted 2023-10-10; First posted 2024-01-18 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Primary Dysmenorrhea
Keywords: Pain; Sacroiliac Joint Dysfunction; Spinal Mobility
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild Primary Dysmenorrhoea: Consists of participants with mild dysmenorrhea according to VAS score
- Moderate Primary Dysmenorrhoea: Consists of participants with moderate dysmenorrhea according to VAS score
- Severe Primary Dysmenorrhoea: Consists of participants with severe dysmenorrhea according to VAS score

SUMMARY:
Evaluation of sacroiliac joint dysfunction in young women with primary dysmenorrhoea using joint provocation and mobility tests and spinal mobility using Spinal Mouse and investigation of the relationship between primary dysmenorrhoea, sacroiliac joint dysfunction and spinal mobility.

DETAILED DESCRIPTION:
Dysmenorrhoea is defined as pathological symptoms associated with menstruation, manifested by abdominal cramps and pain during menstruation and interfering with social life. The pain is of uterine origin and is one of the most common gynaecological disorders in women of childbearing age. It is divided into two types as primary dysmenorrhoea and secondary dysmenorrhoea.

Primary dysmenorrhoea is the most common form and is characterised by cramping pelvic pain that begins shortly before or at the onset of menstruation and lasts for one to three days. It usually begins during puberty and manifests itself with painful menstruation in women with normal pelvic anatomy.

Sacroiliac joint dysfunction is thought to be caused by different causes such as sacroiliac strain, sacroiliac instability and sacroiliac arthritis. One of the distinguishing features is local tenderness in the sacroiliac joint.

There are limited number of studies showing the relationship between sacroiliac joint dysfunction and menstrual cycle. Studies have shown that osteopathic manual therapy techniques applied to the pelvis are effective in alleviating the severity of primary dysmenorrhoea. At the same time, researchers have reported that mobilisation applied to the lumbopelvic regions is good for menstrual pain. Thus, it can be said that mobility is important in primary dysmenorrhoea.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman between the ages of 18-24
* Being single
* Have a regular menstrual cycle (every 24-32 days)
* Duration of menstruation between 3-7 days
* Severity of primary dysmenorrhoea according to VAS

Exclusion Criteria:

* Refusal to participate
* Diagnosis as a patient with secondary dysmenorrhoea
* Presence of chronic disease
* Regular medication
* Polycystic ovary syndrome
* Pelvic inflammatory diseases
* History of uterine, cervical or ovarian cancer
* Previous gynaecological interventions

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Dismonere occurs only in women
Study Population: Only women with a regular menstrual cycle and primary dysmenorrhoea
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Standing Flexion Test | Baseline
  While the patient leans forward with his knees extended, the physiotherapist places his hands behind the patient, just under the spina iliaca posterior superior (SIPS). If one of the SIPS is superior to the other, the test is considered positive.
Sitting Flexion Test | Baseline
  The physical therapist places his fingers just below the bases of the sacrum and just below the angulus inferior lateralis. If any of the SIPS goes more superior than the other, the test is considered positive.
Springing Test | Baseline
  The patient lies in the prone position. While the physiotherapist applies pressure to the sacrum with the hypothenar region of one hand, he tries to detect the posterior sacrum with the other hand.
Gillet Test | Baseline
  The patient is standing. The physiotherapist palpates the SIPS with the thumb of one hand and the sacrum with the other hand. The test is considered positive if there is no or limited postero-inferior movement of the SIPS when the patient flexes the hip-knee.
Hyperextension Test | Baseline
  The patient is standing. The physiotherapist palpates the SIPS with the thumb of one hand and the sacrum with the other hand. The test is considered positive if there is no or limited antero-superior movement of the SIPS when the patient hyperextends the hip.
Gaenslen Test | Baseline
  While the patient lies in the supine position, the physiotherapist passively hangs one of the patient's legs off the bed. In this way, maximum hip hyperextension is achieved. When the other leg is passively flexed, pain in the Sacroiliac Joint (SIJ) on the side hanging from the bed means that the test is positive.
Sacroiliac Compression Test | Baseline
  The patient is positioned in a side-lying position with the knees flexed at 90 degrees and the hips at 45 degrees of flexion. The physiotherapist applies a compression force from the upper iliac crest to the lower iliac crest, and pain in the SIJ means that the test is positive.
Sacroiliac Distraction Test | Baseline
  The patient is positioned supine. The physiotherapist creates distraction force by applying force from the SIPS in the posterior and lateral directions, with his hands crossed. Pain in SIJ means the test is positive.
Posterior Friction Test | Baseline
  The patient is positioned supine. By flexing the hip to 90 degrees and adducting the femur, axial pressure is applied along the femur. Pain over the ilium means the test is positive
Patrick FABER Test | Baseline
  While the patient is in a supine position, his heel is placed on the opposite knee. Thus, flexion, abduction and external rotation movements occur in the hip. The physiotherapist applies force through the opposite side SIPS. The test is considered positive if SIJ pain occurs.

SECONDARY OUTCOMES:
Spinal Mobility Test | Baseline
  Spinal mobility and inclination angle were evaluated using a Spinal Mouse. Spinal Mouse® is a radiation-free device that can measure the curvatures of the spine in the frontal and sagittal planes and transfer it to a computer program via Bluetooth. It can measure 4 different angles: thoracic angle, lumbar angle, inclination angle and sacrum-hip angle.

OTHER OUTCOMES:
Menstruation Symptom Scale (MSS) | Baseline
  It is a five-point Likert-type scale consisting of 24 items. Participants are asked to assign a number between 1 (never) and 5 (always) to the symptoms they experience related to menstruation. The MSS score is calculated by averaging the total score of the items in the scale. An increase in the mean score indicates an increase in the severity of menstrual symptoms.
The Visual Analogue Scale (VAS) | Baseline
  The Visual Analogue Scale (VAS) is the most common scale used to assess pain intensity on a horizontal/vertical bar of 10 or 100 mm. The starting point indicates the absence of pain, while the end point indicates that the pain is too much to bear
Functional and Emotional Dysmenorrhoea (Painful Menstruation) Scale (FEDS) | Baseline
  It is a 5-point Likert-type scale consisting of 14 items. An increase in the mean score indicates an increase in the functional and emotional severity of dysmenorrhoea.The minimum and maximum scores to be obtained from the overall scale are 14 and 70 respectively. As the score increases, the participant's degree of being affected by menstruation increases as well.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Osman PALA, Principal Investigator — Bolu Abant İzzet Baysal University
Locations (1):
- Faculty of Health Sciences Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No